CLINICAL TRIAL: NCT02231086
Title: Adjuvant Hyperthermic Intraperitoneal Chemotherapy in Patients With Colon Cancer at High Risk of Peritoneal Carcinomatosis
Brief Title: Adjuvant HIPEC in High Risk Colon Cancer
Acronym: COLOPEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Health Care Insurance Board (Other)
Responsible Party: Principal Investigator, P.J. Tanis, M.D. Ph.D, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL49960.018.14; 2014-002794-11 (EudraCT Number)
Record Dates: First submitted 2014-08-22; First posted 2014-09-04 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Neoplasms; Peritoneal Neoplasms
Keywords: Chemotherapy, Adjuvant; Laparoscopy; Peritoneal Lavage; HIPEC
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms | interventions — Oxaliplatin; Folfox protocol; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard adjuvant systemic chemotherapy (Active Comparator): Standard adjuvant systemic chemotherapy according to the Dutch colon cancer guideline, using a capecitabine and oxaliplatin (CAPOX) or 5-FU and oxaliplatin (FOLFOX) schedule. Presence or absence of peritoneal recurrence will be evaluated by laparoscopy in case of negative routine examination (CEA and CT thorax/abdomen) at 18 months postoperatively.
  Interventions: Drug: Standard adjuvant systemic chemotherapy; Procedure: Diagnostic laparoscopy
- Adjuvant HIPEC (open/laparoscopic) (Experimental): Adjuvant HIPEC will be performed simultaneously with primary tumor resection, or as a staged procedure (<10 days or 5-8 weeks postoperatively). The chemotherapy during oxaliplatin-HIPEC consists of an intravenous phase with leucovorin 20 mg/m2 (maximum 40 mg) and 5-fluorouracil 400 mg/m2 (maximum 800 mg) and an intraperitoneal phase with oxaliplatin 460 mg/m2 (maximal 920 mg). Standard adjuvant systemic chemotherapy according to the national guideline will be given within 3 weeks from HIPEC. Presence or absence of peritoneal recurrence will be evaluated by laparoscopy in case of negative routine examination (CEA and CT thorax/abdomen) at 18 months postoperatively.
  Interventions: Procedure: Adjuvant HIPEC (open/laparoscopic); Drug: Standard adjuvant systemic chemotherapy; Procedure: Diagnostic laparoscopy

INTERVENTIONS:
Procedure: Adjuvant HIPEC (open/laparoscopic) — Adjuvant HIPEC procedure: access to the abdominal cavity by laparoscopy or laparotomy under general anaesthesia, adhesiolysis if necessary, complete staging of the intra-abdominal cavity, positioning of in- and outflow catheters, perfusion with a minimum of 2l isotonic dialysis fluid at a flow rate of 1-2l/min and an inflow temperature of 42-43˚C. Before the beginning of HIPEC, 5-fluorouracil 400 mg/m2 and leucovorin 20 mg/m2 will be administered intravenously to potentiate oxaliplatin activity. Oxaliplatin (460 mg/m2) is added to the perfusate after attaining at least 42 degrees inflow temperature with a total of 30 minutes perfusion time.
  Other Names: I.V. leucovorin 20 mg/m2 (maximum 40 mg); I.V. 5-fluorouracil 400 mg/m2 (maximum 800 mg); Intraperitoneal oxaliplatin 460 mg/m2 (maximum 920 mg)
  Arms: Adjuvant HIPEC (open/laparoscopic)
Drug: Standard adjuvant systemic chemotherapy — Colon cancer patients with a high risk of developing PC, but do not have (yet) proven macroscopic peritoneal metastasis, are standardly treated with adjuvant systemic chemotherapy. Standard adjuvant systemic chemotherapy consists in the Netherlands of a capecitabine and oxaliplatin (CAPOX) or 5-FU and oxaliplatin (FOLFOX) for a total of 6 months.
  Other Names: adjuvant capecitabine and oxaliplatin (CAPOX); adjuvant 5-FU and oxaliplatin (FOLFOX)
Procedure: Diagnostic laparoscopy — Presence or absence of peritoneal recurrence will be evaluated by laparoscopy in case of negative routine examination (CEA and CT thorax/abdomen) at 18 months postoperatively in both study arms.
  Other Names: Diagnostic laparoscopic surgery

SUMMARY:
This study aims to determine the oncological effectiveness of adjuvant HIPEC, using intraperitoneal oxaliplatin with concomitant i.v. 5-FU/LV, following a curative resection of a T4 or intra-abdominally perforated Colon cancer in preventing the development of peritoneal carcinomatosis in addition to the standard adjuvant systemic treatment.

Hypothesis:

The hypothesis is that adjuvant HIPEC preceding routine adjuvant systemic therapy using i.p. oxaliplatin with concomitant i.v. 5-FU/LV following a curative resection of a T4 or intra-abdominally perforated colon cancer reduces the development of peritoneal carcinomatosis in comparison to standard adjuvant systemic treatment alone.

DETAILED DESCRIPTION:
Background:

The peritoneum is the second most common site of recurrence in patients with colon cancer. Early detection of peritoneal carcinomatosis (PC) by imaging is difficult and adjuvant systemic treatment does not seem to affect peritoneal dissemination in contrast to haematogenous dissemination in the liver or lungs. Of all patients eventually presenting with clinically apparent PC, only a quarter have potentially curable disease. The curative option is cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (CR/HIPEC), but the effectiveness depends highly on the extent of disease and is associated with a considerable complication rate. These clinical problems underline the need for effective adjuvant intraperitoneal therapy in high risk colon cancer patients in order to prevent the development of PC with treatment at a subclinical stage.

Study design:

This will be a multicentre study in which 176 eligible patients will be randomized to adjuvant HIPEC followed by adjuvant systemic chemotherapy in the experimental arm, or the standard adjuvant systemic chemotherapy alone in the control arm. Adjuvant HIPEC will be performed preferably simultaneously or within 10 days after resection of the primary tumour, either by laparoscopy or open approach, similar to the technique used for resection of the primary tumour. If adjuvant HIPEC cannot be performed within 10 days (i.e. complicated postoperative course), the procedure will be delayed until 5 to 8 weeks postoperatively. Subsequently, patients will receive routine adjuvant chemotherapy (CAPOX) within 3 weeks from HIPEC. Diagnostic laparoscopy will be performed routinely after 18 months postoperatively in both arms of the study in patients without evidence of disease based on routine follow-up using CT imaging and CEA. If peritoneal carcinomatosis is found during staging laparoscopy, CR/ HIPEC will be performed in patients with a maximum of 5 involved regions and without evidence of systemic disease.

Study population:

Patients who underwent intentionally curative resection for a T4N0-2M0 or intra-abdominally perforated colon cancer.

Intervention:

Adjuvant HIPEC procedure: access to the abdominal cavity by laparoscopy or laparotomy under general anaesthesia, adhesiolysis if necessary, complete staging of the intra-abdominal cavity, positioning of in- and outflow catheters, perfusion with a minimum of 2l isotonic dialysis fluid at a flow rate of 1-2l/min and an inflow temperature of 42-43˚C. Before the beginning of HIPEC, 5-fluorouracil 400 mg/m2 and leucovorin 20 mg/m2 will be administered intravenously to potentiate oxaliplatin activity. Oxaliplatin (460 mg/m2) is added to the perfusate after attaining at least 42 degrees inflow temperature with a total of 30 minutes perfusion time.

Outcomes:

Primary endpoint is peritoneal recurrence-free survival at 18 months. Secondary endpoints are number of participants with adverse events as a measure of safety and tolerability, incidence of PC at end of follow-up with or without concomitant liver/lung metastases, percentage of false negative CT at 18 months (second look laparoscopy/laparotomy as gold standard), disease-free survival, overall survival, quality of life and costs.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* Intention to start routine adjuvant systemic therapy
* adequate clinical condition to undergo simultaneous HIPEC or re- laparoscopy or re-laparotomy with HIPEC within either 10 days or between week 5-8 from --primary resection
* written informed consent
* white blood cell count of at least 3000/mm3, platelet count of at least 100.000/mm3
* no bleeding diathesis or coagulopathy
* normal creatinine or creatinine clearance of at least 50 ml/min

Exclusion Criteria:

* postoperative complications that interfere with adjuvant HIPEC within 8 weeks (i.e. persisting intra-abdominal abscess, significant fascial dehiscence, enteric fistula)
* no intention to start routine adjuvant systemic therapy
* liver and/or lung metastases
* pregnant or lactating women
* unstable or uncompensated respiratory or cardiac disease
* serious active infections
* other concurrent chemotherapy
* hypersensitivity to fluorouracil, folinic acid or another substance of leucovorin or oxaliplatin
* stomatitis, ulceration in the mouth or gastrointestinal tract.
* severe diarrhea
* severe hepatic and / or renal dysfunction.
* plasma bilirubin concentrations greater than 85 μmol/l.
* pernicious anemia or other anaemias due to vitamin B12 deficiency.
* peripheral sensory neuropathy with functional impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter J. Tanis, M.D., Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (9):
- Netherlands (9):
  - Academic Medical Center, Amsterdam
  - Antoni van Leeuwenhoek hospital, Amsterdam
  - Free University Medical Center, Amsterdam
  - Catharina hospital, Eindhoven
  - University Medical Centre Groningen, Groningen
  - Antonius hospital, Nieuwegein
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Zwanenburg ES, Wisselink DD, Klaver CEL, Bilt JDWV, den Berg JGV, Kodach LL, Nagtegaal ID, Tanis PJ, Snaebjornsson P; COLOPEC collaborators. Underdiagnosis of positive resection margins and synchronous peritoneal metastases in locally advanced colon cancer: histopathological reassessment of primary resection in the COLOPEC trial. Virchows Arch. 2025 Oct;487(4):787-797. doi: 10.1007/s00428-025-04065-x. Epub 2025 May 16. PMID 40374989
- [Derived] Zwanenburg ES, El Klaver C, Wisselink DD, Punt CJA, Snaebjornsson P, Crezee J, Aalbers AGJ, Brandt-Kerkhof ARM, Bremers AJA, Burger PJWA, Fabry HFJ, Ferenschild FTJ, Festen S, van Grevenstein WMU, Hemmer PHJ, de Hingh IHJT, Kok NFM, Kusters M, Musters GD, Schoonderwoerd L, Tuynman JB, van de Ven AWH, van Westreenen HL, Wiezer MJ, Zimmerman DDE, van Zweeden A, Dijkgraaf MGW, Tanis PJ; COLOPEC Collaborators Group; COLOOPEC Collaborators Group. Adjuvant Hyperthermic Intraperitoneal Chemotherapy in Patients With Locally Advanced Colon Cancer (COLOPEC): 5-Year Results of a Randomized Multicenter Trial. J Clin Oncol. 2024 Jan 10;42(2):140-145. doi: 10.1200/JCO.22.02644. Epub 2023 Nov 3. PMID 37922442
- [Derived] Zwanenburg ES, Wisselink DD, Klaver CEL, van der Bilt JDW, Tanis PJ, Snaebjornsson P; COLOPEC trial collaborators. The measured distance between tumor cells and the peritoneal surface predicts the risk of peritoneal metastases and offers an objective means to differentiate between pT3 and pT4a colon cancer. Mod Pathol. 2022 Dec;35(12):1991-2001. doi: 10.1038/s41379-022-01154-z. Epub 2022 Sep 19. PMID 36123540
- [Derived] Klaver CEL, Wisselink DD, Punt CJA, Snaebjornsson P, Crezee J, Aalbers AGJ, Brandt A, Bremers AJA, Burger JWA, Fabry HFJ, Ferenschild F, Festen S, van Grevenstein WMU, Hemmer PHJ, de Hingh IHJT, Kok NFM, Musters GD, Schoonderwoerd L, Tuynman JB, van de Ven AWH, van Westreenen HL, Wiezer MJ, Zimmerman DDE, van Zweeden AA, Dijkgraaf MGW, Tanis PJ; COLOPEC collaborators group. Adjuvant hyperthermic intraperitoneal chemotherapy in patients with locally advanced colon cancer (COLOPEC): a multicentre, open-label, randomised trial. Lancet Gastroenterol Hepatol. 2019 Oct;4(10):761-770. doi: 10.1016/S2468-1253(19)30239-0. Epub 2019 Jul 29. PMID 31371228
- [Derived] Klaver CE, Musters GD, Bemelman WA, Punt CJ, Verwaal VJ, Dijkgraaf MG, Aalbers AG, van der Bilt JD, Boerma D, Bremers AJ, Burger JW, Buskens CJ, Evers P, van Ginkel RJ, van Grevenstein WM, Hemmer PH, de Hingh IH, Lammers LA, van Leeuwen BL, Meijerink WJ, Nienhuijs SW, Pon J, Radema SA, van Ramshorst B, Snaebjornsson P, Tuynman JB, Te Velde EA, Wiezer MJ, de Wilt JH, Tanis PJ. Adjuvant hyperthermic intraperitoneal chemotherapy (HIPEC) in patients with colon cancer at high risk of peritoneal carcinomatosis; the COLOPEC randomized multicentre trial. BMC Cancer. 2015 May 24;15:428. doi: 10.1186/s12885-015-1430-7. PMID 26003804

RESULTS

PARTICIPANT FLOW:
Groups:
- Adjuvant HIPEC (Open/Laparoscopic): Adjuvant HIPEC will be performed simultaneously with primary tumor resection, or as a staged procedure (<10 days or 5-8 weeks postoperatively). The chemotherapy during oxaliplatin-HIPEC consists of an intravenous phase with leucovorin 20 mg/m2 (maximum 40 mg) and 5-fluorouracil 400 mg/m2 (maximum 800 mg) and an intraperitoneal phase with oxaliplatin 460 mg/m2 (maximal 920 mg). Standard adjuvant systemic chemotherapy according to the national guideline will be given within 3 weeks from HIPEC. Presence or absence of peritoneal recurrence will be evaluated by laparoscopy in case of negative routine examination (CEA and CT thorax/abdomen) at 18 months postoperatively.
  Adjuvant HIPEC (open/laparoscopic): Adjuvant HIPEC procedure: access to the abdominal cavity by laparoscopy or laparotomy under general anaesthesia, adhesiolysis if necessary, complete staging of the intra-abdominal cavity, positioning of in- and outflow catheters, perfusion with a minimum of 2l isotonic dialysis fluid
Period: Overall Study
Arm/Group | Standard Adjuvant Systemic Chemotherapy | Adjuvant HIPEC (Open/Laparoscopic)
Started | 102 | 102
Completed | 63 | 65
Not Completed | 39 | 37

BASELINE CHARACTERISTICS:
Population: Intention-to-treat Baseline population
Groups:
- Adjuvant HIPEC (Open/Laparoscopic): Adjuvant HIPEC will be performed simultaneously with primary tumor resection, or as a staged procedure (<10 days or 5-8 weeks postoperatively). The chemotherapy during oxaliplatin-HIPEC consists of an intravenous phase with leucovorin 20 mg/m2 (maximum 40 mg) and 5-fluorouracil 400 mg/m2 (maximum 800 mg) and an intraperitoneal phase with oxaliplatin 460 mg/m2 (maximal 920 mg). Standard adjuvant systemic chemotherapy according to the national guideline will be given within 3 weeks from HIPEC. Presence or absence of peritoneal recurrence will be evaluated by laparoscopy in case of negative routine examination (CEA and CT thorax/abdomen) at 18 months postoperatively.
  Adjuvant HIPEC (open/laparoscopic): Adjuvant HIPEC procedure: access to the abdominal cavity by laparoscopy or laparotomy under general anaesthesia, adhesiolysis if necessary, complete staging of the intra-abdominal cavity, positioning of in- and outflow catheters, perfusion with a minimum of 2l isotonic dialysis flui
- Total: Total of all reporting groups
Arm/Group | Standard Adjuvant Systemic Chemotherapy | Adjuvant HIPEC (Open/Laparoscopic) | Total
Number analyzed (Participants) | 102 | 100 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 67 | 134
  >=65 years | 35 | 33 | 68
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [54 to 68] | 61.5 [56 to 68] | 61 [55 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 97
  Male | 52 | 53 | 105
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Intention-to-treat Baseline population
  Participants
    Netherlands | 102 | 100 | 202

OUTCOME MEASURES:

1. Primary Outcome: Peritoneal Recurrence Free Survival at 18 Months
Description: Peritoneal recurrence-free survival at 18 months determined by CT and CEA. If CEA was normal and CT did not show any signs of peritoneal metastase at 18 months, a diagnostic laparoscopy was performed in those patients who consented to this intervention. Complete peritoneal staging was performed during laparoscopy, and biopsies were taken from suspicious lesions. If no peritoneal lesions were seen or biopsies were negative, this indicated that the patient was free from peritoneal recurrence.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Standard Adjuvant Systemic Chemotherapy | Adjuvant HIPEC (Open/Laparoscopic)
Number analyzed (Participants) | 102 | 100
participants | 79 | 80

2. Secondary Outcome: Treatment Related Toxicity of Adjuvant HIPEC
Description: Toxicity directly related to adjuvant HIPEC included 30-day complication rate, re-intervention rate, and re-admission rate.
Time Frame: 30 days after adjuvant HIPEC
Population: Only measured in experimental group
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Adjuvant Systemic Chemotherapy | Adjuvant HIPEC (Open/Laparoscopic)
Number analyzed (Participants) | 0 | 87
Participants | 0 | 0

3. Secondary Outcome: Hospital Stay for Simultaneous and Staged HIPEC, Either Open or Laparoscopic
Description: Hospital stay for simultaneous and staged HIPEC, either open or laparoscopic.
Time Frame: 10 weeks
Reporting Status: Not Posted

4. Secondary Outcome: False-negative Rate of CT-scan for Peritoneal Metastases
Description: The presence or absence of peritoneal metastasis on CT-scan will be compared to the findings during diagnostic laparoscopy, histological biopsy or fine needle aspiration cytology.
Time Frame: 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Patterns of Dissemination (Peritoneal Plus or Minus Distant Metastases)
Description: Patterns of dissemination (peritoneal plus or minus distant metastases).
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2022-02

6. Secondary Outcome: Disease-free Survival
Description: Disease-free survival.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2022-02

7. Secondary Outcome: Overall Survival
Description: Overall survival.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2022-02

8. Secondary Outcome: Quality of Life Questionnaire Survey 5- Year Follow-up
Description: Quality of life questionnaire survey 5- year follow-up.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2022-02

ADVERSE EVENTS:
Time Frame: All postoperative complications after resection of the primary tumor and after adjuvant HIPEC, as well as adverse events occuring during adjuvant chemotherapy were collected, until 30 days after last trial related intervention, for an average of 2 years.
Description: We used standard definitions for AE and SAE
Arm/Group | Standard Adjuvant Systemic Chemotherapy | Adjuvant HIPEC (Open/Laparoscopic)
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/100
Serious Adverse Events (participants affected / at risk) | 46/102 | 95/100
Other Adverse Events (participants affected / at risk) | 102/102 | 100/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Adjuvant Systemic Chemotherapy (N=102) | Adjuvant HIPEC (Open/Laparoscopic) (N=100)
Anastomotic leakage (Surgical and medical procedures) | 0 | 2
wound infection (Surgical and medical procedures) | 4 | 7
Obstructive ileus (Gastrointestinal disorders) | 1 | 3
Paralytic ileus (Gastrointestinal disorders) | 4 | 5
Gastroparesis (Gastrointestinal disorders) | 8 | 15
abscess (Infections and infestations) | 1 | 3
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
delirium (Nervous system disorders) | 1 | 4
line sepsis (Infections and infestations) | 0 | 1
venous thrombosis (Blood and lymphatic system disorders) | 0 | 1
atrial fibrillation (Cardiac disorders) | 0 | 4
Electrolyte disorder (Metabolism and nutrition disorders) | 6 | 8
parenteral feeding (Metabolism and nutrition disorders) | 9 | 22
dehydration (Renal and urinary disorders) | 1 | 1
colonic stenosis (Surgical and medical procedures) | 0 | 1
cardiopulmonary resuscitation (General disorders) | 1 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
cardiac (Cardiac disorders) | 1 | 2
urologic (Renal and urinary disorders) | 2 | 8
ovarian cyst (Reproductive system and breast disorders) | 1 | 0
gastric perforation (Surgical and medical procedures) | 1 | 0
nodal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
chemical peritonitis (Injury, poisoning and procedural complications) | 1 | 1
encapsulating peritoneal sclerosis (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Adjuvant Systemic Chemotherapy (N=102) | Adjuvant HIPEC (Open/Laparoscopic) (N=100)
diarrhea (Gastrointestinal disorders) | 73 | 68
vomiting (Gastrointestinal disorders) | 24 | 27
peripheral sensible neuropathy (Nervous system disorders) | 73 | 68
mucositis (Gastrointestinal disorders) | 20 | 13
fatigue (General disorders) | 58 | 58
anorexia (Metabolism and nutrition disorders) | 20 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT02231086/Prot_SAP_000.pdf